CLINICAL TRIAL: NCT02842853
Title: Immune Lot Consistency, Immunogenicity, and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Adolescents and Adults Aged 10 to 55 Years
Brief Title: Immune Lot Consistency, Immunogenicity, and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MET43; U1111-1161-3060 (Other: WHO)
Record Dates: First submitted 2016-07-15; First posted 2016-07-25 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; MenACYW Conjugate vaccine; Licensed MCV4 vaccine
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MenACYW Conjugate Vaccine Lot 1 (Experimental): Healthy, meningococcal-vaccine naive adolescents aged 10 to 17 years (Group 1a) and adults aged 18 to 55 years (Group 1b) received a single dose of MenACYW conjugate vaccine from lot 1 on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- MenACYW Conjugate Vaccine Lot 2 (Experimental): Healthy, meningococcal-vaccine naive adolescents aged 10 to 17 years (Group 2a) and adults aged 18 to 55 years (Group 2b) received a single dose of MenACYW conjugate vaccine from lot 2 on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- MenACYW Conjugate Vaccine Lot 3 (Experimental): Healthy, meningococcal-vaccine naive adolescents aged 10 to 17 years (Group 3a) and adults aged 18 to 55 years (Group 3b) received a single dose of MenACYW conjugate vaccine from lot 3 on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Menactra® (Active Comparator): Healthy, meningococcal-vaccine naive adolescents aged 10 to 17 years (Group 4a) and adults aged 18 to 55 years (Group 4b) received a single dose of Menactra® on Day 0.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: MenACYW conjugate vaccine
  Arms: MenACYW Conjugate Vaccine Lot 1; MenACYW Conjugate Vaccine Lot 2; MenACYW Conjugate Vaccine Lot 3
Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra®

SUMMARY:
The purpose of the study was to evaluate immune lot consistency of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine and the immune non-inferiority compared to the licensed vaccine Menactra®, and describe the safety and additional immunogenicity of these study vaccines in adolescents and adults 10 to 55 years of age in the United States (US).

Primary Objectives:

* To demonstrate the immune lot consistency of the antibody responses to meningococcal serogroups A, C, Y, and W following the administration of a single dose of MenACYW Conjugate vaccine with respect to serum bactericidal assay using human complement (hSBA) geometric mean titers (GMTs).
* To demonstrate the non-inferiority of the antibody responses to meningococcal serogroups A, C, Y, and W following the administration of a single dose of MenACYW Conjugate vaccine (pooled Lots 1 to 3) compared to those observed following the administration of a single dose of Menactra®.

Secondary Objective:

* To demonstrate the non-inferiority of the antibody responses to meningococcal serogroups A, C, Y, and W following the administration of a single dose of MenACYW Conjugate vaccine (pooled Lots 1 to 3) compared to those observed following the administration of a single dose of Menactra® in the adult population (18 to 55 years old).
* To demonstrate the non-inferiority of the antibody responses to meningococcal serogroups A, C, Y, and W following the administration of a single dose of MenACYW Conjugate vaccine (pooled Lots 1 to 3) compared to those observed following the administration of a single dose of Menactra® in the adolescent population (10 to 17 years old).
* To compare the hSBA vaccine seroresponses of meningococcal serogroups A, C, Y, and W for each of 3 lots of MenACYW Conjugate vaccine 30 days (+14 days) after vaccination.
* To compare the hSBA antibody GMTs of meningococcal serogroups A, C, Y, and W following the administration of MenACYW Conjugate vaccine to those observed following the administration of Menactra®.

Observational Objectives:

* To describe the safety profile of MenACYW Conjugate vaccine and that of the licensed Menactra®.

DETAILED DESCRIPTION:
Healthy meningococcal-vaccine naïve adolescents and adults were randomized and received a single dose of either MenACYW Conjugate vaccine from 1 of the 3 lots (Lot 1, Lot 2, or Lot 3) or Menactra®. They were assessed for immunogenicity at baseline (pre-vaccination) and at 30 to 44 days post-vaccination. Safety information were collected post-vaccination and throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10 to 55 years on the day of inclusion.
* Informed consent form was signed and dated by the participant (aged 18 to 55 years) or assent form was signed and dated by the participant and informed consent form was signed and dated by the parent(s) or guardian (for participants aged 10 to < 18 years).
* Participant (>= 18 years) or participant (10 to < 18 years) and parent / guardian were able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must have been pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination).
* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which may be received at least 2 weeks before or after the study investigational vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B vaccine).
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Verbal report of thrombocytopenia, as reported by the participant or the participant's parent / guardian, contraindicating intramuscular vaccination in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion.
* Personal history of Guillain-Barre syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine within 10 years of the proposed study vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >= 100.4 degree Fahrenheit [°F]). A prospective participant was not be included in the study until the condition was resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3344 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (75):
- United States (75):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Mobile, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Harrisburg, Arkansas
  - Jonesboro, Arkansas
  - Anaheim, California
  - Downey, California
  - Los Angeles, California
  - Paramount, California
  - Redding, California
  - Sacramento, California
  - San Diego, California
  - Santa Rosa, California
  - Upland, California
  - West Covina, California
  - Littleton, Colorado
  - DeLand, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Savannah, Georgia
  - Meridian, Idaho
  - Council Bluffs, Iowa
  - Lenexa, Kansas
  - Newton, Kansas
  - Park City, Kansas
  - Wichita, Kansas
  - Bardstown, Kentucky
  - Metairie, Louisiana
  - Bridgeton, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Corvallis, Oregon
  - Grants Pass, Oregon
  - Erie, Pennsylvania
  - Hermitage, Pennsylvania
  - McMurray, Pennsylvania
  - Upper Saint Clair, Pennsylvania
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Jackson, Tennessee
  - Nashville, Tennessee
  - Tullahoma, Tennessee
  - Corpus Christi, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Waxahachie, Texas
  - Draper, Utah
  - Layton, Utah
  - Murray, Utah
  - Orem, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - West Jordan, Utah
  - Burke, Virginia
  - Charlottesville, Virginia
  - Midlothian, Virginia
  - Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 90 centers in the United States (US) from 15 July 2016 to 16 August 2016.
Pre-assignment Details: A total of 3344 participants who met all inclusion and none of the exclusion criteria were enrolled and randomized in the study.
Groups:
- MenACYW Conjugate Vaccine Lot 1: Healthy, meningococcal-vaccine naive adolescents aged 10 to 17 years (Group 1a) and adults aged 18 to 55 years (Group 1b) received a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine from lot 1 on Day 0.
Period: Overall Study
Arm/Group | MenACYW Conjugate Vaccine Lot 1 | MenACYW Conjugate Vaccine Lot 2 | MenACYW Conjugate Vaccine Lot 3 | Menactra®
Started | 902 | 895 | 906 | 641
Vaccinated | 895 | 886 | 900 | 636
Safety Analysis Set (SafAS) (SafAS: participants who received at least 1 dose of study vaccine & had any safety data available.) | 895 | 883 | 898 | 635
Completed | 879 | 861 | 885 | 617
Not Completed | 23 | 34 | 21 | 24
Not completed — Non-compliance with the protocol | 3 | 7 | 2 | 5
Not completed — Subject met exclusion criteria | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 13 | 9 | 8
Not completed — Lost to Follow-up | 9 | 13 | 10 | 11

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | MenACYW Conjugate Vaccine Lot 1 | MenACYW Conjugate Vaccine Lot 2 | MenACYW Conjugate Vaccine Lot 3 | Menactra® | Total
Number analyzed (Participants) | 902 | 895 | 906 | 641 | 3344
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 402 | 400 | 397 | 329 | 1528
  Between 18 and 65 years | 500 | 495 | 509 | 312 | 1816
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.4 (15.6) | 27.1 (15.7) | 27.3 (15.5) | 25.6 (15.4) | 27.0 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 535 | 531 | 496 | 357 | 1919
  Male | 367 | 364 | 410 | 284 | 1425
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 191 | 207 | 188 | 141 | 727
  Not Hispanic or Latino | 710 | 685 | 716 | 500 | 2611
  Unknown or Not Reported | 1 | 3 | 2 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 7 | 5 | 3 | 16
  Asian | 9 | 19 | 19 | 14 | 61
  Native Hawaiian or Other Pacific Islander | 6 | 4 | 3 | 2 | 15
  Black or African American | 175 | 186 | 166 | 121 | 648
  White | 680 | 647 | 683 | 478 | 2488
  More than one race | 30 | 29 | 30 | 21 | 110
  Unknown or Not Reported | 1 | 3 | 0 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 902 | 895 | 906 | 641 | 3344

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Meningococcal Serogroups A, C, Y, And W Antibodies Following Vaccination With 3 Lots of MenACYW Conjugate Vaccine
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by serum bactericidal assay using human complement (hSBA). Data for this outcome measure were not planned to be collected and analyzed for the Menactra® reporting group.
Time Frame: Day 30 (post-vaccination)
Population: Per-Protocol Analysis Set (PPAS) defined for accessing ACYW immune response data for participants who received at least one dose of study vaccine & had a valid post-vaccination serology result. Participants who presented pre-defined protocol deviations were excluded. Here, "Number analyzed" = participants with available data for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | MenACYW Conjugate Vaccine Lot 1 | MenACYW Conjugate Vaccine Lot 2 | MenACYW Conjugate Vaccine Lot 3
Number analyzed (Participants) | 843 | 820 | 845
Titer (1/dilution)
  Serogroup A: number analyzed (Participants) | 843 | 819 | 843
  Serogroup A | 84.9 [75.8 to 95.1] | 96.5 [86.4 to 108] | 97.9 [87.7 to 109]
  Serogroup C: number analyzed (Participants) | 841 | 820 | 845
  Serogroup C | 326 [286 to 372] | 305 [267 to 349] | 352 [307 to 405]
  Serogroup Y: number analyzed (Participants) | 843 | 820 | 844
  Serogroup Y | 213 [191 to 238] | 210 [188 to 234] | 218 [194 to 246]
  Serogroup W: number analyzed (Participants) | 843 | 820 | 844
  Serogroup W | 84.5 [75.1 to 95.1] | 81.6 [72.7 to 91.5] | 87.2 [77.2 to 98.5]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 2; Serogroup A: Lot 1 vs Lot 2; Test type: Equivalence — Lot consistency was demonstrated across the 3 lots, if, for each pair of lots and each antigen, the 2-sided 95% Confidence Interval (CI) for the ratio of the GMTs lies between 1/2 and 2; GMT Ratio = 0.880, 95% CI 2-sided [0.751 to 1.03]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine Lot 2 vs MenACYW Conjugate Vaccine Lot 3; Serogroup A: Lot 2 vs Lot 3; Test type: Equivalence — Lot consistency was demonstrated across the 3 lots, if, for each pair of lots and each antigen, the 2-sided 95% CI for the ratio of the GMTs lies between 1/2 and 2; GMT Ratio = 0.985, 95% CI 2-sided [0.843 to 1.15]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 3; Serogroup A: Lot 1 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.867, 95% CI 2-sided [0.740 to 1.02]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 2; Serogroup C: Lot 1 vs Lot 2; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 1.07, 95% CI 2-sided [0.888 to 1.29]
Statistical Analysis 5: Comparison: MenACYW Conjugate Vaccine Lot 2 vs MenACYW Conjugate Vaccine Lot 3; Serogroup C: Lot 2 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.866, 95% CI 2-sided [0.714 to 1.05]
Statistical Analysis 6: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 3; Serogroup C: Lot 1 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.927, 95% CI 2-sided [0.766 to 1.12]
Statistical Analysis 7: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 2; Serogroup Y: Lot 1 vs Lot 2; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 1.02, 95% CI 2-sided [0.869 to 1.19]
Statistical Analysis 8: Comparison: MenACYW Conjugate Vaccine Lot 2 vs MenACYW Conjugate Vaccine Lot 3; Serogroup Y: Lot 2 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.961, 95% CI 2-sided [0.816 to 1.13]
Statistical Analysis 9: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 3; Serogroup Y: Lot 1 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.975, 95% CI 2-sided [0.829 to 1.15]
Statistical Analysis 10: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 2; Serogroup W: Lot 1 vs Lot 2; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 1.04, 95% CI 2-sided [0.878 to 1.22]
Statistical Analysis 11: Comparison: MenACYW Conjugate Vaccine Lot 2 vs MenACYW Conjugate Vaccine Lot 3; Serogroup W: Lot 2 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.936, 95% CI 2-sided [0.791 to 1.11]
Statistical Analysis 12: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 3; Serogroup W: Lot 1 vs Lot 3; Test type: Equivalence — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.970, 95% CI 2-sided [0.818 to 1.15]

2. Primary Outcome: Percentage of Participants Achieving hSBA Vaccine Seroresponse for Meningococcal Serogroups A, C, Y And W Following Vaccination With Either MenACYW Conjugate Vaccine or Menactra® Vaccine
Description: Antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA. The hSBA vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >= 1:16 for participants with pre-vaccination hSBA titers < 1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >= 1:8.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here, "Number analyzed"=participants with available data for specified category. Data for this outcome measure were planned to be analyzed for the pooled population of MenACYW Conjugate vaccine reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled): Healthy, meningococcal-vaccine naive adolescents aged 10 to 17 years and adults aged 18 to 55 years received single dose of MenACYW Conjugate vaccine from any of the lots 1, 2 or 3 on Day 0.
Arm/Group | MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) | Menactra®
Number analyzed (Participants) | 2508 | 593
percentage of participants
  Serogroup A: number analyzed (Participants) | 2503 | 593
  Serogroup A | 73.8 [72.0 to 75.5] | 54.6 [50.5 to 58.7]
  Serogroup C: number analyzed (Participants) | 2503 | 593
  Serogroup C | 88.8 [87.5 to 90.0] | 47.9 [43.8 to 52.0]
  Serogroup Y: number analyzed (Participants) | 2505 | 593
  Serogroup Y | 91.4 [90.3 to 92.5] | 73.4 [69.6 to 76.9]
  Serogroup W: number analyzed (Participants) | 2505 | 593
  Serogroup W | 80.3 [78.7 to 81.8] | 61.2 [57.2 to 65.2]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup A; Test type: Non-Inferiority — 95% CI of the difference was calculated from the Wilson Score Method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference is > -10% for all serogroups; Percentage Difference = 19.1, 95% CI 2-sided [14.8 to 23.5]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup C; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 40.9, 95% CI 2-sided [36.7 to 45]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 18.1, 95% CI 2-sided [14.5 to 21.9]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 19.1, 95% CI 2-sided [14.9 to 23.3]

3. Secondary Outcome: Percentage of Participants Achieving hSBA Vaccine Seroresponse for Meningococcal Serogroups A, C, Y And W Following Vaccination With Either MenACYW Conjugate Vaccine or Menactra® Vaccine in Adults
Description: Antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA. The hSBA vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >= 1:16 for participants with pre-vaccination hSBA titers < 1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >= 1:8. Only adults aged 18-55 years who received a single dose of Menactra® (Group 4b) or MenACYW Conjugate vaccine (Group 1b-3b) from any of the lots 1, 2 or 3, were included in this outcome measure.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here, "Overall number of participants analyzed" = participants evaluable for this outcome measure; and "Number analyzed"= participants with available data for specified category. Data for this outcome measure were planned to be analyzed for the pooled population of MenACYW Conjugate vaccine reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) | Menactra®
Number analyzed (Participants) | 1410 | 293
percentage of participants
  Serogroup A: number analyzed (Participants) | 1406 | 293
  Serogroup A | 73.5 [71.2 to 75.8] | 53.9 [48.0 to 59.7]
  Serogroup C: number analyzed (Participants) | 1406 | 293
  Serogroup C | 83.4 [81.4 to 85.3] | 42.3 [36.6 to 48.2]
  Serogroup Y: number analyzed (Participants) | 1408 | 293
  Serogroup Y | 88.1 [86.3 to 89.8] | 60.8 [54.9 to 66.4]
  Serogroup W: number analyzed (Participants) | 1408 | 293
  Serogroup W | 77.0 [74.7 to 79.2] | 50.2 [44.3 to 56.0]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup A; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 19.6, 95% CI 2-sided [13.5 to 25.8]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup C; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 41.1, 95% CI 2-sided [35.0 to 46.9]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 27.4, 95% CI 2-sided [21.7 to 33.3]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 26.8, 95% CI 2-sided [20.7 to 32.9]

4. Secondary Outcome: Percentage of Participants Achieving hSBA Vaccine Seroresponse for Meningococcal Serogroups A, C, Y And W Following Vaccination With Either MenACYW Conjugate Vaccine or Menactra® Vaccine in Adolescents
Description: Antibody titers against meningococcal serogroups A, C, Y, and W measured by hSBA. The hSBA vaccine seroresponse for serogroups A, C, Y, and W was defined as post-vaccination hSBA titers >= 1:16 for participants with pre-vaccination hSBA titers < 1:8 or at least a 4-fold increase in hSBA titers from pre- to post-vaccination for participants with pre-vaccination hSBA titers >= 1:8. Only adolescents aged 10-17 years who received a single dose of Menactra® (Group 4a) or MenACYW Conjugate vaccine (Group 1a-3a) from any of the lots 1, 2 or 3, were included in this outcome measure.
Time Frame: Day 30 (post-vaccination)
Population: Analysis performed on PPAS. Here, "Overall number of participants analyzed" = participants evaluable for this outcome measure; and "Number analyzed" = participants with available data for specified category. Data for this outcome measure were planned to be analyzed for the pooled population of MenACYW Conjugate vaccine reporting groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) | Menactra®
Number analyzed (Participants) | 1098 | 300
percentage of participants
  Serogroup A: number analyzed (Participants) | 1097 | 300
  Serogroup A | 74.0 [71.3 to 76.6] | 55.3 [49.5 to 61.0]
  Serogroup C: number analyzed (Participants) | 1097 | 300
  Serogroup C | 95.6 [94.2 to 96.8] | 53.3 [47.5 to 59.1]
  Serogroup Y: number analyzed (Participants) | 1097 | 300
  Serogroup Y | 95.6 [94.2 to 96.8] | 85.7 [81.2 to 89.4]
  Serogroup W: number analyzed (Participants) | 1097 | 300
  Serogroup W | 84.5 [82.2 to 86.6] | 72.0 [66.6 to 77.0]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup A; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 18.7, 95% CI 2-sided [12.5 to 24.9]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup C; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 42.3, 95% CI 2-sided [36.6 to 48.0]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 10.0, 95% CI 2-sided [6.18 to 14.5]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage Difference = 12.5, 95% CI 2-sided [7.22 to 18.2]

5. Secondary Outcome: Percentage of Participants Achieving hSBA Vaccine Seroresponse for Meningococcal Serogroups A, C, Y And W Following Vaccination With 3 Lots of MenACYW Conjugate Vaccine
Description: as for outcome 2
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here, "Number analyzed" = participants with available data for specified category. Data for this outcome measure were not planned to be collected and analyzed for the Menactra® reporting group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MenACYW Conjugate Vaccine Lot 1 | MenACYW Conjugate Vaccine Lot 2 | MenACYW Conjugate Vaccine Lot 3
Number analyzed (Participants) | 843 | 820 | 845
percentage of participants
  Serogroup A: number analyzed (Participants) | 842 | 818 | 843
  Serogroup A | 71.1 [67.9 to 74.2] | 76.5 [73.5 to 79.4] | 73.7 [70.6 to 76.6]
  Serogroup C: number analyzed (Participants) | 840 | 819 | 844
  Serogroup C | 90.5 [88.3 to 92.4] | 89.1 [86.8 to 91.2] | 86.7 [84.3 to 88.9]
  Serogroup Y: number analyzed (Participants) | 842 | 819 | 844
  Serogroup Y | 92.4 [90.4 to 94.1] | 91.9 [89.9 to 93.7] | 89.9 [87.7 to 91.9]
  Serogroup W: number analyzed (Participants) | 842 | 819 | 844
  Serogroup W | 81.5 [78.7 to 84.0] | 80.7 [77.8 to 83.4] | 78.7 [75.8 to 81.4]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 2; Serogroup A: Lot 1 vs Lot 2; Test type: Other; Percentage Difference = -5.4, 95% CI 2-sided [-9.59 to -1.16]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine Lot 2 vs MenACYW Conjugate Vaccine Lot 3; Serogroup A: Lot 2 vs Lot 3; Test type: Other; Percentage Difference = 2.9, 95% CI 2-sided [-1.3 to 7.01]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 3; Serogroup A: Lot 1 vs Lot 3; Test type: Other; Percentage Difference = -2.5, 95% CI 2-sided [-6.78 to 1.74]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 2; Serogroup C: Lot 1 vs Lot 2; Test type: Other; Percentage Difference = 1.3, 95% CI 2-sided [-1.58 to 4.28]
Statistical Analysis 5: Comparison: MenACYW Conjugate Vaccine Lot 2 vs MenACYW Conjugate Vaccine Lot 3; Serogroup C: Lot 2 vs Lot 3; Test type: Other; Percentage Difference = 2.4, 95% CI 2-sided [-0.740 to 5.54]
Statistical Analysis 6: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 3; Serogroup C: Lot 1 vs Lot 3; Test type: Other; Percentage Difference = 3.7, 95% CI 2-sided [0.708 to 6.79]
Statistical Analysis 7: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 2; Serogroup Y: Lot 1 vs Lot 2; Test type: Other; Percentage Difference = 0.5, 95% CI 2-sided [-2.14 to 3.07]
Statistical Analysis 8: Comparison: MenACYW Conjugate Vaccine Lot 2 vs MenACYW Conjugate Vaccine Lot 3; Serogroup Y: Lot 2 vs Lot 3; Test type: Other; Percentage Difference = 2.0, 95% CI 2-sided [-0.763 to 4.79]
Statistical Analysis 9: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 3; Serogroup Y: Lot 1 vs Lot 3; Test type: Other; Percentage Difference = 2.5, 95% CI 2-sided [-0.248 to 5.20]
Statistical Analysis 10: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 2; Serogroup W: Lot 1 vs Lot 2; Test type: Other; Percentage Difference = 0.8, 95% CI 2-sided [-3.00 to 4.54]
Statistical Analysis 11: Comparison: MenACYW Conjugate Vaccine Lot 2 vs MenACYW Conjugate Vaccine Lot 3; Serogroup W: Lot 2 vs Lot 3; Test type: Other; Percentage Difference = 2.0, 95% CI 2-sided [-1.84 to 5.89]
Statistical Analysis 12: Comparison: MenACYW Conjugate Vaccine Lot 1 vs MenACYW Conjugate Vaccine Lot 3; Serogroup W: Lot 1 vs Lot 3; Test type: Other; Percentage Difference = 2.8, 95% CI 2-sided [-1.02 to 6.61]

6. Secondary Outcome: Geometric Mean Titers (GMTs) of Meningococcal Serogroups A, C, Y, and W Antibodies Following Vaccination With MenACYW Conjugate and Menactra®
Description: Antibody titers of meningococcal serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis performed on PPAS. Here, "Overall number of participants analyzed" = participants evaluable for this outcome measure; and "Number analyzed"= number of participants with available data for specified category. Data for this outcome measure were planned to be analyzed for the pooled population of MenACYW Conjugate vaccine reporting groups.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Groups:
- MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled): Healthy, meningococcal-vaccine naive adolescents aged 10 to 17 years and adults aged 18 to 55 years received 0.5 mL of MenACYW Conjugate vaccine from any of the lots 1, 2 or 3 on Day 0.
Arm/Group | MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) | Menactra®
Number analyzed (Participants) | 2508 | 593
Titer (1/dilution)
  Serogroup A: number analyzed (Participants) | 2505 | 593
  Serogroup A | 92.9 [87.1 to 99.1] | 48.1 [41.8 to 55.2]
  Serogroup C: number analyzed (Participants) | 2506 | 593
  Serogroup C | 328 [303 to 354] | 40.7 [33.8 to 49.0]
  Serogroup Y: number analyzed (Participants) | 2507 | 593
  Serogroup Y | 214 [200 to 228] | 66.4 [56.4 to 78.0]
  Serogroup W: number analyzed (Participants) | 2507 | 593
  Serogroup W | 84.4 [78.8 to 90.4] | 44.5 [38.3 to 51.7]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup A; Test type: Other; GMT Ratio = 1.93, 95% CI 2-sided [1.67 to 2.24]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup C; Test type: Other; GMT Ratio = 8.05, 95% CI 2-sided [6.58 to 9.84]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup Y; Test type: Other; GMT Ratio = 3.22, 95% CI 2-sided [2.71 to 3.84]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine (Groups 1, 2, 3 Pooled) vs Menactra®; Serogroup W; Test type: Other; GMT Ratio = 1.90, 95% CI 2-sided [1.61 to 2.24]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to 30 days after vaccination. Solicited reaction (SR) data were collected within 7 days after vaccination. Serious adverse event (SAE) data were collected throughout the study (up to 180 days after vaccination).
Description: Analysis was performed on Safety Analysis Set. A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Groups:
- Menactra: Healthy, meningococcal-vaccine naive adolescents aged 10 to 17 years (Group 4a) and adults aged 18 to 55 years (Group 4b) received a single dose of Menactra® on Day 0.
Arm/Group | MenACYW Conjugate Vaccine Lot 1 | MenACYW Conjugate Vaccine Lot 2 | MenACYW Conjugate Vaccine Lot 3 | Menactra
All-Cause Mortality (participants affected / at risk) | 0/895 | 0/883 | 0/898 | 0/635
Serious Adverse Events (participants affected / at risk) | 9/895 | 13/883 | 6/898 | 5/635
Other Adverse Events (participants affected / at risk) | 477/895 | 485/883 | 489/898 | 353/635
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACYW Conjugate Vaccine Lot 1 (N=895) | MenACYW Conjugate Vaccine Lot 2 (N=883) | MenACYW Conjugate Vaccine Lot 3 (N=898) | Menactra (N=635)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Gastrointestinal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Alcoholic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Somatic symptom disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACYW Conjugate Vaccine Lot 1 (N=895) | MenACYW Conjugate Vaccine Lot 2 (N=883) | MenACYW Conjugate Vaccine Lot 3 (N=898) | Menactra (N=635)
Injection site erythema (General disorders) | 45 | 39 | 43 | 25
Injection site pain (General disorders) | 344 | 339 | 333 | 235
Malaise (General disorders) | 184 | 186 | 189 | 132
Myalgia (Musculoskeletal and connective tissue disorders) | 278 | 271 | 294 | 192
Headache (Nervous system disorders) | 247 | 248 | 253 | 175

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT02842853/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT02842853/SAP_001.pdf